CLINICAL TRIAL: NCT04329260
Title: Mutation of the LEPR Gene at Reunion Island: Involvement in Pediatric Obesity GRÉOL (Génétique Réunion Obésité LEPR)
Brief Title: Mutation of the LEPR Gene at Reunion Island: Involvement in Pediatric Obesity
Acronym: GREOL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/CHU/04
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric population: Children between 3 to 18 years old with severe (BMI> IOTF-30) and early (before the age of 6) obesity.
  A Saliva sample for screening of the deletion Δ6-8 of LEPR gene will be performed for each child.
- Adult member family: The screening of the same deletion according the same procedure will be proposed to the adult family member if the child presents the deletion Δ6-8 of LEPR gene.

SUMMARY:
The objective of this study is to estimate the proportion of the recurrent deletion Δ6-8 of the LEPR gene in the homozygous and heterozygous state in pediatric cases with severe and early ( before the age of 6) obesity (BMI ≥ IOTF-30) on Reunion Island.

DETAILED DESCRIPTION:
The study of the deletion Δ6-8 of the LEPR gene starts with a saliva sample using a swab in children aged between 3 to 18 years old.

The DNA from this sample will then be analyzed by the PCR technique. If the deletion of the LEPR gene is confirmed in the patient, his adult family members will also be screened using the same procedure.

ELIGIBILITY:
Inclusion Criteria:

* patient with early severe and non syndromic obesity (BMI> IOTC-30) (before 6 years old)
* adult family members with deletion of LEPR gene
* informed consent form signed by participants or parents
* affiliation to social security scheme

Exclusion Criteria:

* patient with syndromic obesity
* patient Under guardianship or Under judicial protection

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between 3 to 18 years old with severe obesity (BMI>30) and adult family members.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of the Δ6-8 deletion of the LEPR gene in paediatric population | at inclusion
  Presence of the deletion of the LEPR gene

SECONDARY OUTCOMES:
Proportion of the Δ6-8 deletion of the LEPR gene in adult family members | 6 months after inclusion of the paediatric population
  Presence of the deletion of the LEPR gene

CONTACTS AND LOCATIONS:
Overall Officials: Paul GUEGUEN, MD, Principal Investigator — CHU de La Réunion

IPD SHARING:
Plan to Share IPD: No